CLINICAL TRIAL: NCT02745093
Title: The Effectiveness, Safety, and Acceptability of Home-administered Medical Abortion at Gestational Age of 8 to ≤9 Weeks Versus >9 to ≤12 Weeks: A Prospective Cohort Study in Mexico City
Brief Title: Medical Abortion at Gestational Age of 8 to ≤9 Weeks Versus >9 to ≤12 Weeks
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ibis Reproductive Health (Other)
Collaborators: Marie Stopes International (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSI-6103
Record Dates: First submitted 2015-08-07; First posted 2016-04-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Medical Abortion
Keywords: Abortion induced; Patient Acceptance of Healthcare; safety; effectiveness; misoprostol; mifepristone
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 64-84 days gestational age (Experimental): Women whose pregnancies are estimated to have a gestational age of 64-84 days will receive 200 µg mifepristone followed by misoprostol 24-48 hours later.
  Interventions: Drug: Mifepristone; Drug: Misoprostol
- 57-63 days gestational age (No Intervention): Women whose pregnancies are estimated to have a gestational age of 57-63 days. (Women in this arm receive the standard of care for medical termination of pregnancy in the stated gestational age range: 200 µg mifepristone administered orally in the clinic on Day 1 then 800 μg misoprostol administered sublingually 24-48 hours later at home with a subsequent dose of 400 μg misoprostol sublingually 6 hours later if she has not expelled the pregnancy).

INTERVENTIONS:
Drug: Mifepristone — Women at 64-84 days' gestation will use the following dosing regimen: 200 µg mifepristone administered orally in the clinic on Day 1.
  Arms: 64-84 days gestational age
Drug: Misoprostol — The client will then be given a total of 2400 µg misoprostol tablets to take home, and will be instructed to take 800 μg misoprostol administered sublingually 24-48 hours later at home and to administer a subsequent dose of 400 μg misoprostol sublingually every 3 hours up to a total of four further doses or until expulsion of the products of conception, whichever comes first.
  Arms: 64-84 days gestational age

SUMMARY:
The purpose of this study is to assess the effectiveness, safety, and acceptability of home-administered medical abortion at gestational age of 8 to ≤9 weeks versus >9 to ≤12 weeks among a cohort of women in Mexico City.

DETAILED DESCRIPTION:
Medical abortion represents an important alternative to surgical methods for termination of early pregnancy. In Mexico City, abortion is legal on request up to 12 weeks of gestation; however, medical abortion is currently only offered up to 10 weeks at Marie Stopes Mexico clinics. The World Health Organization guidelines state that medical abortion drugs may be used to terminate pregnancy up to a gestational age of 24 weeks in clinical settings, with recommended regimens differing by gestational age. However, data are lacking on the safety and effectiveness of home-based medical abortion regimens for pregnancy terminations between >9 and ≤12 weeks' gestation. Investigators propose a prospective cohort study with women between 8 and ≤9 weeks and >9 and ≤12 weeks of pregnancy at Marie Stopes Mexico clinics to compare the effectiveness, safety, and acceptability of mifepristone followed by home-based misoprostol use in these two gestational age groups. The information from this study will inform policy and practice guidelines in Mexico City and potentially other locations by providing evidence on the safety, effectiveness, and acceptability of home-use of medical abortion between >9 and ≤12 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Intrauterine pregnancy 57- 84 days, assessed using clinical assessment and transvaginal or transabdominal ultrasound by crown-rump length (machines will be calibrated and will use a standardized conversion formula to determine gestational age)
* Eligible for medical abortion according to doctor assessment
* Elected medical abortion over surgical abortion after comprehensive counselling
* Haemoglobin level ≥10 g/dl measured by Hemocue
* Willing and able to sign consent forms
* Able to speak and read Spanish
* Agree to comply with the study procedures and visit schedule
* Access to own telephone and to emergency transportation
* Access to a toilet with privacy
* Reside no more than 30 minutes car journey from the Sta. Mónica Hospital in Polanco or the Marie Stopes Mexico Roma Clinic

Exclusion Criteria:

* History or evidence of disorders that represent a contraindication to the use of mifepristone or misoprostol (chronic adrenal failure, severe asthma uncontrolled by corticosteroid therapy, inherited porphyries, glaucoma, mitral stenosis, hepatic or renal disease)
* History of bleeding disorder or current anticoagulant therapy
* Previous allergic reaction to any drugs in the regimen
* Suspicion of any pathology of pregnancy (e.g. molar, ectopic, non-viable pregnancy)
* Multiple gestation
* Presence of an intrauterine device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with complete abortion without surgical intervention by day 30 from mifepristone administration, regardless of misoprostol dosing, by gestational age group | 2-4 weeks

SECONDARY OUTCOMES:
Experience of any major adverse event overall, and by type (emergency room treatment, hospitalization, transfusion, unrecognized ectopic pregnancy, allergic reaction, infection requiring intravenous treatment, and death), by gestational age group | 2-4 weeks
Proportion of participants by gestational age group with complete abortion without surgical intervention after 1, 2, 3, 4, and 5 doses of misoprostol, by gestational age group | 2-4 weeks
Number of participants requiring surgical intervention to complete an abortion due to an ongoing pregnancy, by gestational age group | 2-4 weeks
Number of participants requiring surgical intervention to complete an abortion due to the presence of a persistent non-viable sac, by gestational age group | 2-4 weeks
Number of participants requiring surgical intervention to complete an abortion due to substantial debris in uterus, by gestational age group | 2-4 weeks
Number of participants requiring surgical intervention to complete an abortion due to excessive prolonged bleeding indicated as severe on the adverse event form, by gestational age group | 2-4 weeks
Number of participants requiring surgical intervention to complete an abortion due to woman's request, by gestational age group | 2-4 weeks
Number of participants requiring an unscheduled clinic visit, by gestational age group | 2-4 weeks
Number of participants who called the helpline, by gestational age group | 2-4 weeks
Time to expulsion in days, by gestational age group | 2-4 weeks
Side effects overall and by type (chills, fever, vomiting, nausea, diarrhoea, and severe pain), by gestational age group | 2-4 weeks
Duration of heavy bleeding, by gestational age group | 2-4 weeks
Duration of work or school missed, by gestational age group | 2-4 weeks
Pain reliever use | 2-4 weeks
Satisfied or very satisfied with abortion method, by gestational age group | 2-4 weeks
Would choose medical abortion again instead of surgical, by gestational age group | 2-4 weeks
Would recommend abortion method to a friend, by gestational age group | 2-4 weeks
Proportion of participants who saw products of pregnancy, by gestational age group | 2-4 weeks
Proportion of participants who saw products of pregnancy who reported feelings as: nothing/no feeling, relieved, sad, uncomfortable, other, by gestational group | 2-4 weeks
Received family planning by follow-up visit, by gestational age group / method type/ pregnancy intention | 2-4 weeks
Know where to get contraceptive supplies in the future, by gestational age group and pregnancy intention | 2-4 weeks
Did not receive a contraceptive method by follow-up visit, but don't want to get pregnant in next 12 months, by gestational age group | 2-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Grossman, MD, Principal Investigator — Ibis Reproductive Health
Locations (3):
- Mexico (3):
  - Marie Stopes Mexico Azcapotzalco, Del. Azcapotzalco, Mexico Distrito Federal
  - Marie Stopes Mexico Roma, Del. Cuauhtémoc, Mexico Distrito Federal
  - Marie Stopes Mexico Pedregal, Del. Tlalpan, Mexico Distrito Federal

REFERENCES:
- [Background] Boersma AA, Meyboom-de Jong B, Kleiverda G. Mifepristone followed by home administration of buccal misoprostol for medical abortion up to 70 days of amenorrhoea in a general practice in Curacao. Eur J Contracept Reprod Health Care. 2011 Apr;16(2):61-6. doi: 10.3109/13625187.2011.555568. Epub 2011 Feb 9. PMID 21303309
- [Background] Chen MJ, Creinin MD. Mifepristone With Buccal Misoprostol for Medical Abortion: A Systematic Review. Obstet Gynecol. 2015 Jul;126(1):12-21. doi: 10.1097/AOG.0000000000000897. PMID 26241251
- [Background] Gomperts R, van der Vleuten K, Jelinska K, da Costa CV, Gemzell-Danielsson K, Kleiverda G. Provision of medical abortion using telemedicine in Brazil. Contraception. 2014 Feb;89(2):129-33. doi: 10.1016/j.contraception.2013.11.005. Epub 2013 Nov 12. PMID 24314910
- [Background] Gouk EV, Lincoln K, Khair A, Haslock J, Knight J, Cruickshank DJ. Medical termination of pregnancy at 63 to 83 days gestation. Br J Obstet Gynaecol. 1999 Jun;106(6):535-9. doi: 10.1111/j.1471-0528.1999.tb08320.x. PMID 10426609
- [Background] Hamoda H, Ashok PW, Flett GM, Templeton A. Medical abortion at 9-13 weeks' gestation: a review of 1076 consecutive cases. Contraception. 2005 May;71(5):327-32. doi: 10.1016/j.contraception.2004.10.015. PMID 15854631
- [Background] Hamoda H, Ashok PW, Flett GM, Templeton A. A randomised controlled trial of mifepristone in combination with misoprostol administered sublingually or vaginally for medical abortion up to 13 weeks of gestation. BJOG. 2005 Aug;112(8):1102-8. doi: 10.1111/j.1471-0528.2005.00638.x. PMID 16045525
- [Background] Kulier R, Kapp N, Gulmezoglu AM, Hofmeyr GJ, Cheng L, Campana A. Medical methods for first trimester abortion. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD002855. doi: 10.1002/14651858.CD002855.pub4. PMID 22071804
- [Background] Ngo TD, Park MH, Shakur H, Free C. Comparative effectiveness, safety and acceptability of medical abortion at home and in a clinic: a systematic review. Bull World Health Organ. 2011 May 1;89(5):360-70. doi: 10.2471/BLT.10.084046. Epub 2011 Mar 4. PMID 21556304
- [Background] Safe Abortion: Technical and Policy Guidance for Health Systems. 2nd edition. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK138196/ PMID 23700650
- [Background] Winikoff B, Dzuba IG, Chong E, Goldberg AB, Lichtenberg ES, Ball C, Dean G, Sacks D, Crowden WA, Swica Y. Extending outpatient medical abortion services through 70 days of gestational age. Obstet Gynecol. 2012 Nov;120(5):1070-6. doi: 10.1097/aog.0b013e31826c315f. PMID 23090524